CLINICAL TRIAL: NCT02098278
Title: A Phase 2 Pilot Study to Assess the Safety and Efficacy of CAT-2003 in Patients With Chylomicronemia
Brief Title: Pilot Study To Assess CAT-2003 in Patients With Chylomicronemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CAT-2003-203
Record Dates: First submitted 2014-03-24; First posted 2014-03-28 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Lipoprotein Lipase Deficiency, Familial; Hyperlipoproteinemia Type I; Chylomicronemia, Familial; Hypertriglyceridemia
MeSH Terms: conditions — Hyperlipoproteinemia Type I; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAT-2003 or Placebo (Experimental): All patients will receive placebo for 1 week, and CAT-2003 for 12 weeks during the 13 week treatment period.
  Interventions: Drug: CAT-2003; Drug: Placebo

INTERVENTIONS:
Drug: CAT-2003
Drug: Placebo

SUMMARY:
The purpose of this study is to assess safety and efficacy of CAT-2003 in patients with chylomicronemia. The study will evaluate the effects of CAT-2003 on fasting total and chylomicron triglyceride levels, as well as postprandial total and chylomicron triglyceride clearance.

This is a single-blind study. All patients will receive placebo for 1 week, and CAT-2003 for 12 weeks during the 13 week treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Familial Chylomicronemia (Fasting triglycerides ≥ 880 mg/dL at Screening and documented history of plasma post-heparin LDL activity < 20% of normal or genetic confirmation of homozygosity or compound heterozygosity for loss-of-function mutations in familial chylomicronemia-causing genes) OR
* Non-familial Chylomicronemia (Fasting triglycerides ≥ 440 mg/dL at Screening and documented history of fasting triglycerides ≥ 880 mg/dL)

Key Exclusion Criteria:

* History of any major cardiovascular event within 6 months of Screening
* Type I diabetes mellitus or use of insulin
* History of pancreatitis within 3 month of Screening

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in fasting triglycerides in patients with chylomicronemia | 12 Weeks

SECONDARY OUTCOMES:
Absolute and percent change from baseline on postprandial total and chylomicron triglyceride levels | 12 Weeks
Absolute and percent change from baseline on chylomicron triglyceride clearance | 12 Weeks
Absolute and percent change from baseline in plasma non-HDL-C | 12 Weeks
Frequency of adverse events | 13 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Chicoutimi, Quebec
  - Québec, Quebec